CLINICAL TRIAL: NCT06749704
Title: Effect of High Protein Diet on Hepatic Steatosis, Inflammation and Mitochondrial Bioenergetics in Patients With MAFLD : A Randomized Controlled Trial
Brief Title: Effect of High Protein Diet on Hepatic Steatosis in Patients With MAFLD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-MAFLD-01
Record Dates: First submitted 2024-05-06; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-05

CONDITIONS: Metabolic Dysfunction Associated Fatty Liver Disease
Keywords: mitochondrial dysfunction; metabolic inflexibility; FGF21 resistance
MeSH Terms: conditions — Mitochondrial Diseases | interventions — Diet, High-Protein

STUDY DESIGN:
Intervention Model Description: Open Label
Masking Description: As it is a nutritional intervention study masking either the participant or the investigator is not possible
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Treatment Group (Active Comparator): The intervention is planned as a supervised dietary supplementation, with a goal of restricting the calorie intake to 20 Kcal/Kg BW/day, with a protein intake of 0.9 gm/Kg BW/day i.e., around 15 % of total calories from protein, 25% from fats and 60% from carbohydrates.
  Physical activity recommendations: Brisk walking on a treadmill (at a speed 5-6 Kmph for 60 minutes) OR 5000 steps per day by pedometer counting.
  Interventions: Dietary Supplement: Normal Protein diet
- High Protein Diet (Experimental): The intervention is planned as a supervised dietary supplementation, with a goal of restricting the calorie intake to 20 Kcal/Kg BW/day, with a protein intake of 1.3 gm/Kg BW/day i.e., around 25 % of total calories from protein, 25% from fats and 50% from carbohydrates. Major portion of the protein would be met by dairy, legumes and pulses along with egg whites.
  Physical activity recommendations: Brisk walking on a treadmill (at a speed 5-6 Kmph for 60 minutes) OR 5000 steps per day by pedometer counting.
  Interventions: Dietary Supplement: High protein diet

INTERVENTIONS:
Dietary Supplement: High protein diet — High protein diet
  Arms: High Protein Diet
Dietary Supplement: Normal Protein diet — Normal protein diet
  Arms: Standard Treatment Group

SUMMARY:
MAFLD is a growing problem in India. Its pathophysiology is complex, but focused on abnormal substrate handling due to mitochondrial dysfunction reflecting as metabolic inflexibility. Nutrition is the cornerstone of management. The ideal macronutrient distribution within a hypocaloric diet is not known yet. Evidence from experimental and a few human studies in obese, highlight the role of dietary proteins, independent of calorie restriction, in reducing hepatic steatosis by improving the cellular and systemic bioenergetics.

DETAILED DESCRIPTION:
Novelty: First study to assess the effect of high protein diet (HPD) in comparison to a standard protein diet (SPD) within a calorie restricted diet, on both the cellular and systemic bioenergetics in patients with MAFLD.

Objectives: Aims to see the effect of HPD on hepatic steatosis, cellular and systemic bioenergetics, along with metabolic parameters in patients with MAFLD.

Method: In this RCT, patients with MAFLD (n=140) with or without MS, would be randomized into HPD or SPD groups (i.e. 70 in each group), and parameters like hepatic steatosis (CAP by Transient elastography (FibroScan), cellular bioenergetics by oxygen consumption rate (OCR) and extracellular acidification rate (ECAR) as measured using Seahorse Analyzer, and Indirect Calorimetry will be used to assess the fasting and postglucose challenge (Oral glucose tolerance test) REE and RQ. DEXA scan would be used to assess body composition apart from routine blood tests to assess features of Metabolic syndrome. The serum levels of GLP1, CKK, Ghrelin, FGF21, Adipokines like leptin and adiponectin, NADH/NAD ratio, insulin and glucagon would be measured.

Outcome: A HPD is expected to improve hepatic steatosis, blunted fuel switching (RQ) and cellular bioenergetics (OCR) along with metabolic parameters in patients with MAFLD.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed treatment naïve consenting adults with MAFLD (controlled attenuation parameter; CAP >250, BMI>23 and/or DM) Age 18-65 years

Exclusion Criteria:

* • Lean (BMI <23) patients

  * Age <18 and >65 years
  * Individuals who had been hospitalized with complications of Diabetes mellitus, Chronic Kidney disease, Hypertension in the previous 6 months
  * Patients with viral hepatitis
  * Patients with significant alcohol consumption (regular consumption of > 10g per day for females and > 20g/d in males),
  * Patients having chronic inflammatory bowel disease or any chronic and autoimmune diseases will be excluded
  * Pregnant & lactating women

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-12-27 (Estimated); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of Hepatic steatosis. | 3 months
  Changes in hepatic steatosis at baseline and follow up would be done using fibro scan (CAP) and Computed Tomography (Liver Attenuation Index).

SECONDARY OUTCOMES:
Assessment of cellular bioenergetics would be done. | 3 months
  Changes in oxygen consumption rate (OCR in pmol/min) at baseline and follow up would be done using Seahorse XF analyser.
Assessment of cellular bioenergetics would be done. | 3 months
  Changes in Extracellular acidification rate(ECAR in mph/min) at baseline and follow up would be done using Seahorse XF analyser.
Assessment of systemic bioenergetics would be done. | 3 months
  A switch in Respiratory quotient (RQ) at fasting and OGTT would be assessed using indirect calorimetry at baseline and follow up.
Assessment of metabolic markers at baseline and follow up. | 3 months
  Changes in metabolic markers would be done at baseline and follow up. The following metabolic markers would be assessed :- Blood pressure(systolic and dystolic), HbA1c,Thyroid stimulating hormone , Total lipid profile, CRP levels.
Assessment of muscle mass. | 3 months
  Assessment of muscle mass would be done by DEXA scan at baseline and follow up.
Assessment of serum levels of FGF21(in ng/ml) and leptin(in ng/ml). | 3 months
  Assessments would be done using commercially available Elisa kits at baseline and follow up.
Assessment of serum levels of adiponectin(in μg/mL). | 3 months
  Assessments would be done using commercially available Elisa kits at baseline and follow up.
Assessment of serum levels of insulin(in μU/mL) | 3 months
  Assessments would be done using commercially available Elisa kits at baseline and follow up.
Assessment of serum levels of glucagon(in pg/mL). | 3 months
  Assessments would be done using commercially available Elisa kits at baseline and follow up.
Assessment of serum levels of glucagon like peptide(GLP-1) (in pmol/L) | 3 months
  Assessments would be done using commercially available Elisa kits at baseline and follow up.
Assessment of serum levels of ghrelin (in fmol/ml). | 3 months
  Assessments would be done using commercially available Elisa kits at baseline and follow up.
Assessment of serum levels of cholecystokinin (in pmol/liter). | 3 months
  Assessments would be done using commercially available Elisa kits at baseline and follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Jaya Benjamin, PhD, Study Director — Institute of Liver and Biliary Sciences
Locations (1):
- Institute of Liver and Biliary Sciences, Delhi, New Delhi, India